CLINICAL TRIAL: NCT05909267
Title: Effects of Pharmacological Dopamine Modulation on Motivation and Motor Function in Major Depression Characterized by Low-grade Inflammation.
Brief Title: Dopamine Modulation of Motivation and Motor Function in Major Depression & Inflammation
Acronym: MOTIVADE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Prof. Dr. Stefan M. Gold (Unknown); Prof. Dr. Soyoung Q Park (Unknown); Dr. Ulrike Grittner (Unknown); Motognosis GmbH (Unknown)
Responsible Party: Principal Investigator, Woo Ri Chae, MD, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: MOTIVADE
Record Dates: First submitted 2023-05-31; First posted 2023-06-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Depressive Disorder, Major
Keywords: depression; inflammation; anhedonia; psychomotor retardation
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Inflammation; Anhedonia; Psychomotor Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-dopa/Carbidopa followed by placebo (Experimental): Participants will receive first L-dopa/Carbidopa (100/25 mg), and then placebo.
  Interventions: Drug: L-dopa/Carbidopa; Drug: Placebo
- Placebo followed by L-dopa/Carbidopa (Experimental): Participants will receive first placebo, and then L-dopa/Carbidopa (100/25 mg).
  Interventions: Drug: L-dopa/Carbidopa; Drug: Placebo

INTERVENTIONS:
Drug: L-dopa/Carbidopa — Patients and healthy controls will receive one time administration of L-dopa/Carbidopa (100/25 mg).
Drug: Placebo — Patients and healthy controls will receive one time administration of Placebo.

SUMMARY:
A large body of evidence on depression heterogeneity point to an "immunometabolic" subtype characterized by the clustering of immunometabolic dysregulations with atypical behavioral symptoms related to energy homeostasis. Motivational and motor impairments reflected by symptoms of anhedonia and psychomotor retardation in major depression are closely related to alterations in energy homeostasis, are associated with increased inflammation, and may be a direct consequence of the impact of inflammatory cytokines on the dopamine system in the brain. In the proposed project, the investigators will examine the effect of dopamine stimulation on motivation and motor function in patients with major depression and healthy controls and the role of inflammation using a double-blind, randomized, placebo-controlled, cross-over design. If successful, this study would provide crucial evidence that pharmacologic strategies that increase dopamine may effectively treat inflammation-related symptoms of anhedonia and psychomotor retardation in major depression.

ELIGIBILITY:
Inclusion Criteria:

For patients with major depressive disorder:

* diagnosis of major depressive disorder according to DSM-5
* free of antidepressant medication

For healthy participants:

* C-reactive protein (CRP): ≤ 1 mg/l
* free of antidepressant medication
* free of any current psychiatric disorder

Exclusion Criteria:

* diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, dementia, and current/past alcohol or drug dependence
* central nervous system diseases
* neurological diseases
* suspicious undiagnosed skin lesions or a history of melanoma
* narrow-angle or wide-angle glaucoma
* bronchial asthma
* history of peptic ulcer disease
* history of seizures
* any severe somatic disease
* current infections or chronic inflammatory diseases (e.g., rheumatic diseases, inflammatory bowel disease)
* pregnancy / breast-feeding
* class 3 obesity (body mass index of 40 or higher)
* Use of medication containing reserpine (certain antihypertensive agents), tricyclic antidepressants, bon-selective monoamine oxidase (MAO) inhibitors, antiparkinsonian drugs, sympathomimetic drugs, tetrabenazine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The change in response bias (logb) after L-dopa/Carbidopa compared to placebo in the Probabilistic Reward Task (PRT). | All participants will be tested on two separate experimental sessions separated by an interval of 48 hours, after L-dopa/Carbidopa or placebo.
  The PRT, which uses a signal detection paradigm, will be used to measure response bias, the propensity to select the more rewarded response ("rich").
The change in mean gait speed [m/s] after L-dopa/Carbidopa compared to placebo in the dual task. | All participants will be tested on two separate experimental sessions separated by an interval of 48 hours, after L-dopa/Carbidopa or placebo.
  The dual task mean gait speed will be measured with six wearable inertial measurement units. In this dual task, participants walk at their usual speed while naming as many animals as possible.

SECONDARY OUTCOMES:
The change in choice of the hard task after L-dopa/Carbidopa compared to placebo in the Effort Expenditure for Rewards Task (EEfRT). | All participants will be tested on two separate experimental sessions separated by an interval of 48 hours, after L-dopa/Carbidopa or placebo.
  The EEfRT, a widely used, multi-trial task in which participants are given an opportunity on each trial to choose between two different task difficulty levels in order to obtain monetary rewards, will be used as an objective measure of reward motivation. The EEfRT is reported as the percent of high effort (hard) trials selected. A higher percentage reflects higher motivation for effort expenditure.
The change in movement time [ms] after L-dopa/Carbidopa compared to placebo in the Reaction Time Task (RTI). | All participants will be tested on two separate experimental sessions separated by an interval of 48 hours, after L-dopa/Carbidopa or placebo.
  The RTI from the Cambridge Neuropsychological Test Automated Battery (CANTAB) will be used to assess movement time, which is the time taken to touch the stimulus on the computer screen after the press pad had been released.
The change in risk propensity after L-dopa/Carbidopa compared to placebo in the Risky Decision-Making Task. | All participants will be tested on two separate experimental sessions separated by an interval of 48 hours, after L-dopa/Carbidopa or placebo.
  In the Risky Decision-Making Task, participants have to make choices between a risky option and a safe alternative. Risk Propensity, the proportion of risk-taking trials, will be a secondary outcome.
Response bias (logb) in the PRT | After administration of placebo on Day 2 or Day 3.
Mean gait speed [m/s] in the dual task | After administration of placebo on Day 2 or Day 3.
Choice of the hard task in the EEfRT | After administration of placebo on Day 2 or Day 3.
Movement time [ms] in the RTI | After administration of placebo on Day 2 or Day 3.

OTHER OUTCOMES:
The change in speed and accuracy after L-dopa/Carbidopa compared to placebo in the Rapid Visual Information Processing Task (RVP). | All participants will be tested on two separate experimental sessions separated by an interval of 48 hours, after L-dopa/Carbidopa or placebo.
  The RVP from the Cambridge Neuropsychological Test Automated Battery (CANTAB) will be used to assess performance speed (mean latency for correct responses) and accuracy (target sensitivity score).
Risk propensity in the Risky Decision-Making Task | At baseline on Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Woo Ri Chae, MD MSc, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Klinik für Psychiatrie und Psychotherapie, Steglitz, Germany

IPD SHARING:
Plan to Share IPD: Undecided